CLINICAL TRIAL: NCT07144683
Title: Risk Factors for Anastomotic Leakage After Colorectal Surgery.
Brief Title: Anastomotic Leakage After Colorectal Surgery.
Acronym: AL
Status: Recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Other Study IDs: 1607/07/2025
Record Dates: First submitted 2025-08-14; First posted 2025-08-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Anastomotic Leak; Colorectal Cancer; Diverticulitis
Keywords: Anastomotic leakage; Colorectal surgery; Risk factors; Postoperative complications; Predictive model
MeSH Terms: conditions — Anastomotic Leak; Colorectal Neoplasms; Diverticulitis; Postoperative Complications | interventions — Anastomosis, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Undergoing Colorectal Resection with Anastomosis: All eligible patients undergoing elective/emergency colorectal surgery with primary anastomosis (e.g., ileocolic, colocolic, colorectal, or coloanal). Risk factors and outcomes will be monitored prospectively.
  Interventions: Procedure: Patients Undergoing Colorectal Resection with Anastomosis

INTERVENTIONS:
Procedure: Patients Undergoing Colorectal Resection with Anastomosis — All eligible patients undergoing elective/emergency colorectal surgery with primary anastomosis (e.g., ileocolic, colocolic, colorectal, or coloanal)

SUMMARY:
Anastomotic leakage (AL) is a severe complication after colorectal surgery, with incidence rates of 2-30%. This prospective, single-center observational cohort study aims to identify and quantify independent risk factors for AL, determine its incidence and impact on outcomes, and develop a predictive model. Approximately 430 patients undergoing colorectal resection with anastomosis will be enrolled from August 2025 to August 2026. Risk factors will be assessed preoperatively, intraoperatively, and postoperatively. AL will be defined and graded per the International Study Group of Rectal Cancer (ISGRC) criteria.

DETAILED DESCRIPTION:
Anastomotic leakage (AL) remains a major complication after colorectal surgery, contributing to morbidity, mortality, prolonged hospital stays, and increased costs. Its etiology is multifactorial, involving patient, disease, and surgical factors. This study will prospectively evaluate risk factors in a single-center setting to minimize variability.

AL definition (per ISGRC): Defect at anastomotic site causing communication between intra/extraluminal compartments and luminal tract, diagnosed via clinical signs (e.g., peritonitis, fecal discharge), radiological evidence (e.g., CT showing extraluminal air/contrast or fluid collection), or operative verification.

Severity grading:

* Grade A: Asymptomatic/mild, no active treatment.
* Grade B: Requires intervention (e.g., drainage, antibiotics) but no reoperation.
* Grade C: Requires reoperation.

Risk factors categorized as:

* Preoperative: Demographics (age, sex, BMI), comorbidities (ASA score, diabetes, etc.), lifestyle (smoking, alcohol), nutritional status (albumin, CRP), neoadjuvant therapy, medications, diagnosis (e.g., cancer, tumor location), and bowel preparation.
* Intraoperative: Approach (open/laparoscopic), resection type, anastomosis details (hand-sewn/stapled, level, perfusion assessment), peritoneal soiling, diverting stoma, operative time, blood loss/transfusion, drainage, surgeon experience, complications.
* Postoperative: AL diagnosis/severity/management, inflammatory response (CRP, WBC), anemia, complications (ileus, infection), hospital stay, nutritional support, mobilization, reoperation, ICU stay, mortality, pain management.Early detection of leak using inflammatory markers either in the serum or drain fluid. Drain fluid inflammatory markers (Drain Fluid Calprotectin(CP), Drain Fluid C-Reactive Protein (CRP), Drain Fluid Procalcitonin)and Serum inflammatory markers(Serum C-Reactive Protein (CRP), Serum Procalcitonin (PCT), Serum Lactate dehydrogenase (LDH)).

Data from electronic records, surgical notes, nursing charts, and follow-up. Statistical analysis includes descriptive stats, univariate/multivariate logistic regression for risk factors, subgroup analyses, and predictive model development/validation.

The study adheres to the Helsinki Declaration and Good Clinical Practice (GCP). Informed consent is required.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Undergoing elective or emergency colorectal resection with primary anastomosis (e.g., ileocolic, colocolic, colorectal, coloanal)
* Providing written informed consent

Exclusion Criteria:

* Colorectal resection without anastomosis (e.g., end stoma)
* Inflammatory bowel disease (Crohn's, ulcerative colitis)
* History of previous colorectal surgery involving anastomosis
* Pregnancy
* Unable to provide informed consent or comply with follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients undergoing elective/emergency colorectal surgery with primary anastomosis (e.g., ileocolic, colocolic, colorectal, coloanal). No intervention; observational only. Risk factors and outcomes will be monitored prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Anastomotic Leakage (AL) | Within 30 days post-surgery.
  Proportion of patients developing AL within 30 days post-surgery or during hospital stay (whichever longer), diagnosed clinically, radiologically, or operatively per ISGRC definition

SECONDARY OUTCOMES:
Severity of Anastomotic Leakage | Within 30 days post-surgery
  Graded as A (asymptomatic/mild, no treatment), B (requires intervention, no reoperation), or C (requires reoperation) per ISGRC.
Reoperation Rate Due to AL | Within 30 days post-surgery
  Proportion of patients requiring reoperation for AL.
Readmission Rate Due to AL | Within 30 days post-surgery
  Proportion of patients readmitted for AL-related issues.
Length of Hospital Stay | Within 30 days post-surgery.
  Duration of hospitalization (days) for patients with vs. without AL.
Mortality Rate | Within 30 days post-surgery.
  30-day and in-hospital mortality.
Need for Permanent Stoma | Within 90 days post-surgery
  Proportion of patients requiring permanent stoma due to AL.

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Minia University Hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No